CLINICAL TRIAL: NCT05301062
Title: China Radium-223 Safety and Effectiveness stuDy In Real World mCRPC paTients
Brief Title: A Research Called CREDIT Studies How Safe the Study Treatment Radium-223 is and How Well it Works in Chinese Men With Advanced Prostate Cancer That Has Spread to the Bones and Does Not Respond to Treatments for Lowering Testosterone Levels
Acronym: CREDIT
Status: Terminated | Type: Observational
Why Stopped: Due to the changes of standard of care, the slow recruitment of participants, and the similar safety profile data on real-world use of Radium-223 in China has been published.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21720
Record Dates: First submitted 2022-03-21; First posted 2022-03-29 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Castration-resistant Prostate Cancer; Bone Metastases
MeSH Terms: interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radium-223 dichloride treatment: Castration-resistant prostate cancer (CRPC) patients with bone metastases for whom a decision has been made independently by the treating physician and the patient to treat with Radium-223.
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Treatment with Radium-223 should follow the approved local product information according to National Medical Products Administration (NMPA) approved label

SUMMARY:
This is an observational study in which data from Chinese men with metastatic castration-resistant prostate cancer that has spread to the bones and who start Radium-223 therapy is studied.

When tumors form in the prostate, male hormones like testosterone will cause the spread and growth of tumors. Men with prostate cancer can have hormonal or surgical treatment that lowers testosterone. But this may not stop the cancer from growing or spreading in some men. When the prostate cancer is no longer responding to therapies aimed at lowering testosterone (castration resistant) and has spread to the bones (metastatic), it is referred to as bone metastatic castration-resistant prostate cancer.

The study treatment, Radium-223 (also called Xofigo), gives off radiation that helps to kill cancer cells. It is already approved to be used for men whose prostate cancer has spread to the bone with symptoms, but not to be used for other types of tumors or for prostate cancer that has spread to other parts of the body. Sometimes, after the approval of some drugs, researchers will further study the safety of such approved treatments in patients being treated in routine clinical practice.

In this study, researchers want to learn more about the medical problems that may occur in Chinese patients after they start Radium-223 therapy, especially those problems concerning the blood and blood-forming organs. To answer this question, the researchers will observe patients who start Radium-223 as part of their routine care and also collect information of any medical problems happening after Radium-223 injections from the medical records of these patients. These medical problems may or may not be related to Radium-223 and are also known as adverse events.

The researchers will assess the percentage of men who developed medical problems concerning the blood and blood-forming organs from the start of Radium-223 injection till up to 6 months after the last Radium-223 injection.

The researchers will also collect data on the time the participants live after start of treatment, the change in pain severity, and the time between the end of Radium-223 treatment and the beginning of the following therapy against the cancer.

Besides the data collection, no further tests or examinations of any patients or any samples are planned in this study. The participants will start Radium-223 treatment as part of their routine care as prescribed by their doctors according to the recommended use. Data collection of each participant will last until the participant leaves the study or until the study ends. The study is planned to end 6 months after the last included participant receives the last injection of Radium-223.

ELIGIBILITY:
Inclusion Criteria:

* Male patient
* Histologically or cytologically confirmed castration resistant adenocarcinoma of the prostate with bone metastases
* No visceral metastases
* Decision to initiate treatment with Radium-223 was made independently prior to patient enrollment in the study as per investigator's routine treatment practice
* Signed informed consent

Exclusion Criteria:

* Patients previously treated with Radium-223 for any reason
* Patients currently treated in any other clinical trials including other Radium-223 studies
* Patients are planned for the systemic concomitant use of other radiopharmaceuticals for treatment of prostate cancer or for other use
* Participation in an investigational program with interventions outside of routine clinical practice
* Patients previously treated with Docetaxel
* Patients under treatment with Abiraterone Acetate and the Corticosteroids Prednisone or Prednisolone

Besides Inclusion and exclusion criteria, sites should also follow the locally approved Radium-223 product information

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of CRPC patients with bone metastases treated with Radium-223. Treating physicians (medical oncologists, urologists, nuclear medicine physicians) or designated medical persons will collect historic records and on-study data from the medical records, routine measurements (e.g. tumor assessment). Radium-223 administering physicians in certain circumstances may also collect information including dosing data and other related data from similar sources.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of hematological adverse events | From the start of administration of Radium-223 till up to 6 months after the last Radium-223 administration
  Hematological adverse events are reported as bone marrow suppression

SECONDARY OUTCOMES:
Incidence of other treatment-emergent Adverse events (AEs) and Serious Adverse Events (SAEs) | From the start of administration of Radium-223 till up to 30 days after the last Radium-223 administration
Overall Survival (OS) | From the start of administration of Radium-223 till patient death due to any causes. Up to 30 months
Change in pain severity | From the start of administration of Radium-223 till up to 6 months after the last Radium-223 administration
  Pain severity will be measured using the worst pain score from the Brief pain inventory short form (BPI-SF) questionnaire. The BPI-SF is a self-administered questionnaire with 11 items designed to evaluate the intensity of, and the impairment caused by pain. Four items measure pain intensity using 0 ("no pain") to 10 ("pain as bad as you can imagine") numeric rating scales, and 7 items measure the level of interference with function caused by pain using 0 (no interference) to 10 (complete interference) rating scales.
Time interval from the last administration of Radium-223 to the initiation date of next anti-cancer therapy | From the last administration of Radium-223 till up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, China

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/